CLINICAL TRIAL: NCT03165019
Title: Time Course and Prognostic Significance of Pulmonary Artery Pressure in Highlanders.
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01-8/433
Record Dates: First submitted 2017-05-22; First posted 2017-05-24 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: High Altitude Pulmonary Hypertension; Sleep Apnea
Keywords: high altitude illness; pulmonary hypertension; sleep apnea; disease progression; hypoxia
MeSH Terms: conditions — Pulmonary edema of mountaineers; Sleep Apnea Syndromes; Hypertension, Pulmonary; Disease Progression; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High altitude pulmonary hypertension: Highlanders with high altitude pulmonary hypertension living above 2500 m.
- High altitude control: Healthy highlanders living above 2500 m.
- Low altitude control: Healthy lowlanders living below 1000 m.

SUMMARY:
The purpose of the current study is to evaluate the clinical and physiologic course of Kyrgyz highlanders with high altitude pulmonary hypertension (HAPH) by performing a longitudinal cohort study. To this end, the investigators will invite the same highlanders who participated in the study in 2012 to undergo follow-up examinations in 2017, in order to allow comparisons of current results with baseline data from 2012.

ELIGIBILITY:
Inclusion Criteria:

* high altitude pulmonary hypertension confirmed by clinical presentation and mean pulmonary artery pressure >30 mmHg measured by echocardiography at altitude of residence.
* healthy subjects (high altitude controls)
* Both genders
* Age >16 y
* Kyrgyz ethnicity
* born, raised and currently living at >2500 m
* healthy subjects currently living at <1000 m (low altitude controls)

Exclusion Criteria:

* Pulmonary hypertension from other causes, in particular from left ventricular failure as judged clinically and by echocardiography
* Excessive erythrocytosis
* Other coexistent disorders that may interfere with the cardio-respiratory system and sleep
* Regular use of medication that affects control of breathing
* Heavy smoking

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Highlanders with high altitude pumonary hypertension living at an altitude of 2500-4000 m; healthy highlanders living at an altitude of 2500-4000 m; healthy lowlanders living at an altitude of <1000 m.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Changes in pulmonary artery pressure | Year 2012 to 2017
  Difference in the change in mean pulmonary artery pressure (mPAP measured by echocardiography) 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander

SECONDARY OUTCOMES:
Changes in nocturnal arterial oxygen saturation | Year 2012 to 2017
  Difference in the change in the nocturnal arterial oxygen saturation 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Survival | Year 2012 to 2017
  Cumulative incidence of death and relocation to lower altitudes between 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Progression of oxygen desaturation index | Year 2012 to 2017
  Difference in the change in the oxygen desaturation index 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Progression of quality of life | Year 2012 to 2017
  Difference in the change in the mental and physical component score of the SF-36 questionnaire 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Progression of cognitive performance | Year 2012 to 2017
  Difference in the change in the mean reaction time 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Exercise performance | Year 2012 to 2017
  Difference in the change in 6 minute walk distance 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Arterial blood gas analysis | Year 2012 to 2017
  Difference in the change in arterial blood gases 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander

CONTACTS AND LOCATIONS:
Overall Officials: Talant M Sooronbaev, MD, Principal Investigator — NCCIM
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided